CLINICAL TRIAL: NCT06458257
Title: The Efficacy of Allogeneic Hematopoietic Stem Cell Transplantation in Newly Diagnosed High-relapse-risk CEBPA Mutant Acute Myeloid Leukemia
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shen yang, Chief physician, Ruijin Hospital
Other Study IDs: CEBPA-AML01
Record Dates: First submitted 2024-01-09; First posted 2024-06-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: newly diagnosed; high-relapse-risk; CEBPA mutant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow; peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- HSCT-group: patients received allogeneic hematopoietic stem cell transplantation after consolidation treatment
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation
- Chemo-group: patients received chemotherapy after consolidation treatment
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Allogeneic Hematopoietic Stem Cell Transplantation
  Groups: HSCT-group
Drug: Chemotherapy — Chemotherapy
  Groups: Chemo-group

SUMMARY:
For newly diagnosed high-relapse-risk CEBPA mutant acute myeloid leukemia patients, we aim to perform allogeneic hematopoietic stem cell transplantation after patients finished one cycle of induction and two cycles of consolidation. To access whether the therapeutic regimen is effective for high-relapse-risk CEBPA mutant acute myeloid leukemia, the disease-free-survival (DFS), overall survival (OS), non-relapse-mortality of patients is evaluated.

DETAILED DESCRIPTION:
High-relapse-risk definition:

Participants with non-bZIP in-frame mutations, WT1 mutated status or CD7 negative status are considered of high-relapse-risk; The positive threshold for flow cytometry MRD was 0.0001%; The MRD threshold of molecular biology is the lowest value of the detection protocol of the center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed CEBPA mutant AML. Diagnostic criteria include the presence of CEBPA mutant gene detected at the molecular level;
2. Patients with high-risk molecular markers or gene mutations, or complex karyotypes for disease recurrence, or flow cytometry/gene MRD positivity after two chemotherapy treatments; high-risk molecular markers or gene mutations include: CD7 positive, WT1 mutation, non-bzip-inframe CEBPA mutation; The positive threshold for flow cytometry MRD was 0.0001%; The MRD threshold of molecular biology is the lowest value of the detection protocol of the center.
3. Medical history and diagnosis of MICM, exclusion of MDS, transformation and treatment-related AML;
4. Age 18-65 years old (18 years old ≤Age< 65 years old);
5. Liver and kidney function: blood bilirubin ≤ 35 μmol/L, AST/ALT below 2 times the upper limit of normal, serum creatinine ≤ 150 μmol/L;
6. Normal cardiac function (EF≥50%, New York Cardiac Function Classification NYHA I/II);
7. Physical condition score 0-2 (ECOG score);
8. For patients with peripheral blood leukocytes < 50*109/L at the initial onset, no chemotherapy has been given except for hydroxyurea before the start of induction therapy;
9. For patients with peripheral blood leukocytes ≥ 50*109/L at the initial onset, cytarabine and hydroxyurea are allowed to be treated before the start of induction therapy;
10. Non-pregnant and lactating women;
11. For all women of childbearing age, a pregnancy test must be performed to measure hCG to rule out pregnancy;
12. Obtain informed consent signed by the patient or family member.

Exclusion Criteria:

1. MDS-converted AML, treatment-related AML; mixed cell leukemia; AML patients with central nervous system infiltrates and extramedullary lesions at the time of onset;
2. Relapse patients;
3. Allergies or contraindications to any of the drugs involved in the protocol;
4. Liver and kidney function are obviously abnormal, exceeding the enrollment criteria;
5. Cardiac disease: including echocardiogram EF <50%, cardiac insufficiency (New York cardiac function classification NYHA: III/IV), pericardial effusion (CTCAE score >2) within six months after acute myocardial infarction, ECG QTc >470ms;
6. Lung diseases: pulmonary edema, pleural effusion (CTCAE score >2);
7. Suffering from malignant tumors of other organs at the same time;
8. Active patients with HAV, HBV, HCV and tuberculosis, HIV-positive patients;
9. Concomitant other hematologic diseases (including coagulation abnormalities unrelated to leukemia);
10. Inability to understand or follow the study protocol;
11. Those who participate in other clinical studies at the same time; Presence of any other condition that would preclude the conduct of the study

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosed in Ruijin Hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
disease-free-survival | from data of AML diagnosis until the data of AML relapse, assessed up to 3 years
  disease-free-survival
The relation of CEBPA Mutant AML genetics subgroup with MRD negativity rate after chemotherapy and DFS after transplantation | from enrollment to study completion, a maximum of 3 years
  The relation of CEBPA Mutant AML genetics subgroup with MRD negativity rate after chemotherapy and DFS after transplantation

SECONDARY OUTCOMES:
non-relapse-mortality | from enrollment to study completion, a maximum of 3 years
  non-relapse-mortality
overall survival | from enrollment to study completion, a maximum of 3 years
  overall survival
adverse events | from enrollment to study completion, a maximum of 3 years
  adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes